CLINICAL TRIAL: NCT07137078
Title: Pilates Versus Gyrotonic Expansion System on Chemotherapy Induced Peripheral Neuropathy and Fall Risk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Ahmed Abd El hady El Fahl,ph.d, Assisstant professor, MTI University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005944
Record Dates: First submitted 2025-08-16; First posted 2025-08-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Neuropathy
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (Pilates exercise (Experimental): Pilates exercises, particularly those focusing on core stability, balance, and flexibility, are highly beneficial for individuals at risk of falls. These exercises enhance proprioception, which is the body's ability to sense movement, action, and location, thereby improving coordination and balance. For example, exercises like the "Single Leg Stretch" and "Roll-Up" target the abdominal muscles, which are crucial for maintaining stability. Additionally, "Leg Circles" and "Side Planks" help strengthen hip abductors and stabilizers, contributing to better postural alignment and reducing the likelihood of falls. By regularly incorporating Pilates into a fitness routine, individuals can build strength and confidence, ultimately helping to prevent falls and maintain independence.
  Interventions: Other: pilates
- gyrotonic expansion exercise (Experimental): Exercise phase Training Time Warm-Up Gentle, dynamic stretches focusing on the spine, hips, and legs. Gently roll the head from side to side to release tension, Move shoulders in a circular motion to loosen muscles, While standing, rotate the torso gently from side to side, Rotate each ankle in both directions to improve mobility. 5 minutes Core Activation Using pulley rope system the Arch and Curl, to engage the abdominal muscles, Focus on maintaining proper alignment and breathing deeply. 13 minutes Balance and Coordination Using pulley rope system Standing Series, shifting weight, such as the Spiral Sequence, to improve coordination. 12 minutes Flexibility and Range of Motion Leg stretches using the Leg Extension Unit to improve hip and knee range of motion. 5 minutes
  Interventions: Other: gyrotonic expansion exercise
- control (No Intervention): No traninig

INTERVENTIONS:
Other: pilates — Pilates exercises, particularly those focusing on core stability, balance, and flexibility, are highly beneficial for individuals at risk of falls. These exercises enhance proprioception, which is the body's ability to sense movement, action, and location, thereby improving coordination and balance. For example, exercises like the "Single Leg Stretch" and "Roll-Up" target the abdominal muscles, which are crucial for maintaining stability. Additionally, "Leg Circles" and "Side Planks" help strengthen hip abductors and stabilizers, contributing to better postural alignment and reducing the likelihood of falls. By regularly incorporating Pilates into a fitness routine, individuals can build strength and confidence, ultimately helping to prevent falls and maintain independence.
  Arms: (Pilates exercise
Other: gyrotonic expansion exercise — Exercise phase Training Time Warm-Up Gentle, dynamic stretches focusing on the spine, hips, and legs. Gently roll the head from side to side to release tension, Move shoulders in a circular motion to loosen muscles, While standing, rotate the torso gently from side to side, Rotate each ankle in both directions to improve mobility. 5 minutes Core Activation Using pulley rope system the Arch and Curl, to engage the abdominal muscles, Focus on maintaining proper alignment and breathing deeply. 13 minutes Balance and Coordination Using pulley rope system Standing Series, shifting weight, such as the Spiral Sequence, to improve coordination. 12 minutes Flexibility and Range of Motion Leg stretches using the Leg Extension Unit to improve hip and knee range of motion. 5 minutes
  Arms: gyrotonic expansion exercise

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a common and dose-limiting side effect of neurotoxic chemotherapy (ie, taxanes, vinca alkaloids, platinum, and bortezomib) that interferes with patients' daily function and worsens quality of life (1-3). In a study of 512 cancer survivors, 47% reported persistent neuropathy up to 6 years after chemotherapy completion. Furthermore, these survivors exhibited altered gait patterns with slower and shorter steps, as well as a fall risk 1.8-fold greater than that of those without CIPN (4). In another study, 12% of cancer survivors with CIPN reported falls within a 3-month period (5). These evidences highlight the need for an effective treatment for CIPN to improve quality of life and safety among cancer survivors. Current empirical treatments for CIPN include symptom management with analgesics, antidepressants, and antiepileptics (6). However, these approaches are limited not only by toxicities but also by patients' reluctance to further medicate a medication-related condition.

DETAILED DESCRIPTION:
Pilates can be an effective intervention to address patients received chemotherapy and the associated increased risk of falls. CIPN is a common side effect of certain chemotherapy drugs, characterized by nerve damage that leads to symptoms such as pain, tingling, numbness, and weakness primarily in the hands and feet. These symptoms significantly impact balance and mobility, increasing the risk of falls. Pilates, with its focus on core strength, balance, flexibility, and controlled movement, can help mitigate these effects. The slow, deliberate movements in Pilates improve proprioception and strengthen the core and lower extremities, which are crucial for maintaining balance and stability. Regular Pilates practice can enhance postural alignment and muscle coordination, which can reduce the risk of falls in individuals experiencing CIPN.

Pilates can be an effective intervention to address chemotherapy-induced peripheral neuropathy (CIPN) and the associated increased risk of falls. CIPN is a common side effect of certain chemotherapy drugs, characterized by nerve damage that leads to symptoms such as pain, tingling, numbness, and weakness primarily in the hands and feet. These symptoms significantly impact balance and mobility, increasing the risk of falls. Pilates, with its focus on core strength, balance, flexibility, and controlled movement, can help mitigate these effects. The slow, deliberate movements in Pilates improve proprioception and strengthen the core and lower extremities, which are crucial for maintaining balance and stability. Regular Pilates practice can enhance postural alignment and muscle coordination, which can reduce the risk of falls in individuals experiencing CIPN.

The Gyrotonic Expansion System (GES) is an innovative movement methodology that is gaining attention for its potential benefits in addressing chemotherapy side effects, result in numbness, tingling, and pain in the extremities, significantly affecting balance and increasing fall risk. The GES involves fluid, spiraling movements designed to enhance flexibility, strength, coordination, and balance. By promoting increased circulation and nerve stimulation, these movements may help alleviate the symptoms of chemotherapy, potentially improving patient outcomes. The system's focus on core strength and alignment can also aid in stabilizing posture, thereby reducing the likelihood of falls.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* Diagnosed with CIPN
* Completed at least 3 cycles of chemotherapy
* Ability to provide informed consent

Exclusion Criteria:

* Severe neuropathy requiring pharmacological intervention
* Concurrent participation in another physical therapy regimen
* Any medical condition contraindicating physical exercise.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-05 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy Induced Peripheral Neuropathy Assessment Tool | at baseline and at 12 weeks
  The CIPNAT is a fifty item instrument that contains two sets of items symptom experience items and interference items. The 36 symptom experience items measure severity, distress, and frequency of nine neuropathic symptoms including; numbness in the hands, numbness in the feet, tingling in the hands, tingling in the feet, sensitivity to cold temperatures, nerve pain, muscle/joint aches, muscle weakness and loss of balance. Participants are first asked whether they have developed any of the nine symptoms since receiving chemotherapy. For each symptom reported, participants are asked to rate the intensity, distress, and frequency of that symptom on a 0-10 numeric rating scale. The symptom experience item set is scored by adding the number of symptoms reported (0-9) with the severity, distress, and frequency scores for each reported symptom. Scores range from 0-279 with higher scores corresponding with higher levels of CIPN.

SECONDARY OUTCOMES:
Grip Strength | at baseline and at 12 weeks
  Grip strength will be assessed using a Jamar handheld dynamometer.
Dynamic Balance | at baseline and at 12 weeks
  The Four-Square Step Test (FSST) assesses dynamic balance and fall risk. Scores are interpreted based on the time it takes to complete the sequence, with higher scores indicating a greater risk of falls.
Dual Task (DT) Gait Speed | at baseline and at 12 weeks
  The DT gait speed was conducted similarly to the ST gait speed, with the addition of a cognitive task. There are 2 categories of DT commonly used: mental tracking and verbal fluency. Mental tracking tasks require one to hold information in the mind while performing a mental process, and are commonly used to examine sustained attention, information processing speed, and executive function.21 Verbal fluency tasks require spontaneous word production under specific search conditions and are also thought to examine executive function.21 there are currently no established standards for DT gait assessment. Existing literature advises DT selection based on the tested cohort, taking into consideration background diseases and other socio-demographics such as education level.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy ,Cairo University, Cairo, Egypt